CLINICAL TRIAL: NCT06742996
Title: A Phase 3 Randomized Double-Blind Multicenter Study of Sonrotoclax Plus Zanubrutinib Versus Placebo Plus Zanubrutinib in Patients With Relapsed/Refractory Mantle Cell Lymphoma
Brief Title: A Study to Investigate the Efficacy and Safety of Sonrotoclax Plus Zanubrutinib Compared With Placebo Plus Zanubrutinib in Adults With Relapsed/Refractory Mantle Cell Lymphoma (CELESTIAL-RRMCL)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BeOne Medicines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BGB-11417-302; 2024-515593-27-00 (EU CTIS Number); CTR20250207 (Registry Identifier: ChinaDrugTrials)
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Mantle Cell Lymphoma; B Cell Lymphoma
Keywords: mantle cell lymphoma; MCL; relapsed/refractory mantle cell lymphoma; sonrotoclax; BGB-11417
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma, B-Cell | interventions — zanubrutinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: sonrotoclax plus zanubrutinib (Experimental): Sonrotoclax and zanubrutinib will be administered in combination.
  Interventions: Drug: Sonrotoclax; Drug: Zanubrutinib
- Arm B: placebo plus zanubrutinib (Placebo Comparator): Placebo and zanubrutinib will be administered in combination.
  Interventions: Drug: Zanubrutinib; Drug: Placebo

INTERVENTIONS:
Drug: Sonrotoclax — Administered orally
  Other Names: BGB-11417
  Arms: Arm A: sonrotoclax plus zanubrutinib
Drug: Zanubrutinib — Administered orally
  Other Names: Brukinsa; BGB-3111
Drug: Placebo — Administered orally
  Arms: Arm B: placebo plus zanubrutinib

SUMMARY:
The goal of this study is to compare how well sonrotoclax plus zanubrutinib works versus zanubrutinib plus placebo in treating adults with relapsed/refractory (R/R) mantle cell lymphoma (MCL). This study will also look at the safety of sonrotoclax plus zanubrutinib versus zanubrutinib plus placebo.

DETAILED DESCRIPTION:
Our company, previously known as BeiGene, is now officially BeOne Medicines. Because some of our older studies were sponsored under the name BeiGene, you may see both names used for this study on this website.

ELIGIBILITY:
Inclusion Criteria:

* Histologically locally confirmed diagnosis of MCL based on the World Health Organization 2022 classification of Haematolymphoid Tumors (WHO-HAEM5), or based on International Consensus Classification (ICC)
* Ability to provide archival or fresh tumor tissue for retrospective central confirmation of MCL diagnosis
* Received 1 to 5 prior lines of systemic therapy including an anti-CD20 monoclonal antibody (mAb)-based immunotherapy or chemoimmunotherapy and requiring treatment in the opinion of the investigator
* Relapsed or refractory disease after the last line of therapy
* Measurable disease defined as ≥ 1 nodal lesion that is > 1.5 cm in longest diameter, or ≥ 1 extranodal lesion that is > 1 cm in longest diameter
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2
* Adequate organ function

Exclusion Criteria:

* Prior therapy with B-cell lymphoma-2 inhibitor (BCL2i)
* Prior therapy with BTK degraders
* Prior therapy with covalent or non-covalent Bruton tyrosine kinase inhibitor (BTKi) unless the participant was intolerant of non-zanubrutinib covalent or non-covalent BTKi. Participants with refractory disease to BTKi therapy or relapse attributed to failure of BTKi therapy are ineligible.
* Prior autologous stem cell transplantation or chimeric antigen receptor T-cell therapy within 3 months before first dose of study drug
* Prior allogeneic stem cell transplant within 6 months of the first dose of the study drug
* Known central nervous system involvement by lymphoma
* Clinically significant cardiovascular disease
* History of stroke or intracranial hemorrhage within 6 months before first dose of study drug

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2032-03-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) as assessed by Blinded Independent Review Committee (BIRC) | Approximately 41 months
  PFS is defined as the time from randomization to the date of progression or death, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | Approximately 92 months
  OS is defined as the time from randomization to the date of death from any cause.
PFS as assessed by investigator (INV) | Approximately 58 months
  PFS is defined as the time from randomization to the date of progression or death, whichever occurs first.
Overall Response Rate (ORR) as assessed by BIRC and by INV | Approximately 58 months
  ORR is defined as the percentage of participants who achieved a best overall response of partial response (PR) or complete response (CR), per Lugano 2014 criteria.
Duration of Response (DOR) as assessed by BIRC and by INV | Approximately 58 months
  DOR is defined as the time from the first qualifying response to the date of progression or death, whichever occurs first.
Complete Response Rate (CRR) as assessed by BIRC and by INV | Approximately 58 months
  CRR is defined as the percentage of participants who achieved a best overall response of CR.
Time to first response as assessed by BIRC and by INV | Approximately 58 months
  Time to first response is defined as time from the date of randomization to first response.
Time to initiation of new anticancer therapy | Approximately 58 months
  Time to initiation of new anticancer therapy is defined as time from the date of randomization to the date of initiation of new anticancer therapy.
Health-Related Quality of Life (HRQoL) as Assessed by the European Organisation of Research and Treatment of Cancer-Quality of Life Questionnaire Non-Hodgkin Lymphoma High Grade Module 29 (EORTC-QLQ-NHL-HG29) | Approximately 58 months
  Patient-reported symptom burden, neuropathy, and physical condition/fatigue as measured by the EORTC-QLQ-NHL-HG29 questionnaire. The EORTC-QLQ-NHL-HG29 is the NHL-aggressive module of QLQ-C30; and it consists of 5 scales: Symptom burden due to disease and/or treatment (7 items), Neuropathy (2 items), Physical condition/Fatigue (5 items), Emotional impacts (4 items), and Worries/Fears health and functioning (11 items). Items are rated using a 4-point response scale ("not at all," "a little," "quite a bit," and "very much"). A higher score for all the multi-item scales and items represents a higher level of symptomatology or problems.
Health-Related Quality of Life (HRQoL) as Assessed by the European Organisation of Research and Treatment of Cancer-Quality of Life Questionnaire Core 30 (EORTC-QLQ-C30) | Approximately 58 months
  Patient-reported global health status (GHS), role, and physical function as measured by the EORTC-QLQ-C30 questionnaire. The EORTC QLQ-30 contains 30 questions that incorporate 5 functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning), 1 global health status scale, 3 symptom scales (fatigue, nausea and vomiting, and pain), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The participant answers questions about their health during the past week. There are 28 questions answered on a 4-point scale where 1 =Not at all (best) to 4 =Very Much (worst) and 2 questions answered on a 7-point scale where 1 =Very poor (worst) to 7 =Excellent (best).
Number of participants with treatment-emergent adverse events (TEAEs) | From the first dose of study drug(s) to 30 days after the last dose; up to approximately 58 months
  Number of participants with TEAEs, including laboratory values, vital signs, electrocardiogram results, and physical examination findings, graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeOne Medicines
Locations (149):
- United States (35):
  - University of Alabama At Birmingham Hospital, Birmingham, Alabama
  - Mayo Clinic Phoenix, Phoenix, Arizona
  - Yale University, Yale Cancer Center, New Haven, Connecticut
  - Memorial Cancer Institute, Memorial Healthcare System, Pembroke Pines, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Mission Cancer and Blood, Waukee, Iowa
  - University of Maryland Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Dana Farber Cancer Institute Longwood Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - The Cancer and Hematology Centers, Grand Rapids, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Hattiesburg Hematology and Oncology Clinic, Hattiesburg, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Cancer Specialists St Francis Grand Island, Grand Island, Nebraska
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - The Valley Hospital, Inc, Paramus, New Jersey
  - Atrium Health Levine Cancer Institute (Lci), Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - University Hospitals, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Ohio Health Research Institute, Columbus, Ohio
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - McGlinn Cancer Institute, West Reading, Pennsylvania
  - Tennesse Oncology Chattanooga Downtown, Chattanooga, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Md Anderson Cancer Center, Houston, Texas
  - Texas Oncology Austin Midtown, Round Rock, Texas
  - University of Virginia, Charlottesville, Virginia
  - Virgina Cancer Specialists, Gainesville, Virginia
  - Vcu Massey Cancer Center, Richmond, Virginia
  - Northwest Cancer Specialist, Pc(Us Oncology Research), Vancouver, Washington
- Argentina (4):
  - Hospital Aleman, CABA
  - FUNDALEU, Caba
  - Hospital Italiano de Buenos Aires, Ciudad Autonoma Buenos Aires
  - Hospital Universitario de Cordoba, Córdoba
- Australia (10):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Genesiscare North Shore, St Leonards, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Sunshine Coast Hospital and Health Service, Birtinya, Queensland
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Health, Clayton, Victoria
  - Rockingham Hospital, Cooloongup, Western Australia
  - Linear Clinical Research, Nedlands, Western Australia
  - One Clinical Research, Nedlands, Western Australia
  - Perth Blood Institute, West Perth, Western Australia
- Austria (4):
  - Ordensklinikum Linz Gmbh Elisabethinen, Linz
  - Universitatsklinik Fur Innere Medizin Iii Universitatsklinikum Der Pmu Landeskrankenhaus Salzburg, Salzburg
  - Uk St Poelten, Sankt Pölten
  - Medical University Vienna Oncology, Vienna
- Brazil (10):
  - Fundacao Pio Xii Hospital de Amor de Barretos, Barretos
  - Hospital Felicio Rocho, Belo Horizonte
  - Universidade de Campinas Centro de Hematologia E Hemoterapia, Campinas
  - Hospital Erasto Gaertner, Curitiba
  - Instituto Joinvilense de Hematologia E Oncologia, Joinville
  - Fundacao Universidade de Caxias Do Sul Instituto de Pesquisas Em Saude, Petrópolis
  - Hospital de Clinicas de Porto Alegre, Porto AlegreRS
  - Hospital Do Cancer de Pernambuco, Recife
  - Hcfmusp Servico de Hematologia, Hemoterapia E Terapia Celular, São Paulo
  - Hospital Santa Rita de Cassia Afecc, Vitória
- China (21):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Sun Yat Sen University Cancer Center, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Jiangxi Province Cancer Hospital, Nanchang, Jiangxi
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - Shaanxi Provincial Peoples Hospital, Xi'an, Shaanxi
  - Linyi Cancer Hospital, Linyi, Shandong
  - The Affiliated Hospital of Qingdao University Branch West Coast, Qingdao, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Sichuan Academy of Medical Sciences and Sichuan Provincial Peoples Hospital, Chengdu, Sichuan
  - The First Affiliated Hospital, Zhejiang University School of Medicinechengzhan, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
- France (4):
  - Chu Montpellier Hopital Saint Eloi, Montpellier
  - Centre Hospitalier Universitaire Nantes Hotel Dieu, Nantes
  - Chu Hopital Lyon Sud, PierreBenite
  - Chu Tours Hopital Bretonneau, Tours
- Germany (6):
  - Klinikum Chemnitz Ggmbh, Chemnitz
  - Klinikum Der Johann Wolfgang Goethe Universitat, Frankfurt am Main
  - Universitatsklinikum Halle, Halle
  - Universitatsklinikum Hamburg Eppendorf, Hamburg
  - Stauferklinikum Schwabisch Gmund Kliniken Ostalb, Mutlangen
  - Dept of Medicine Iii, University Hospitallmu, München
- Italy (5):
  - Policlinico Sorsola Malpighi, Aou Di Bologna, Bologna
  - Ospedale Vito Fazzi, Asl Lecce, Leece
  - Istituto Romagnolo Per Lo Studio Dei Tumori Dino Amadori Irst, Meldola
  - Azienda Sanitaria Universitaria Giuliano Isontina, Trieste
  - Centroricerche Cliniche Di Verona Srl, Verona
- Japan (18):
  - Aichi Cancer Center Hospital Clinical Oncology, Nagoya, Aichi-ken
  - Toyohashi Municipal Hospital, Toyohashishi, Aichi-ken
  - Chiba Cancer Center, Chiba, Chiba
  - Matsuyama Red Cross Hospital, Matsuyama, Ehime
  - Ogaki Municipal Hospital, Ōgaki, Gifu
  - Hiroshima Red Cross Hospital and Atomic Bomb Survivors Hospital, Hiroshima, Hiroshima
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kobe City Medical Center General Hospital, KobeShi, Hyōgo
  - Kagoshima University Hospital, Kagoshima, Kagoshima-ken
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Tohoku University Hospital, Sendai, Miyagi
  - Kurashiki Central Hospital, Kurashikishi, Okayama-ken
  - Osaka Red Cross Hospital, Osakashi, Osaka
  - Dokkyo Medical University Saitama Medical Center, Koshigaya, Saitama
  - Institute of Science Tokyo Hospital, Bunkyoku, Tokyo
  - National Hospital Organization Okayama Medical Center, Okayama
  - Osaka Metropolitan University Hospital, Osaka
  - Yokohama Municipal Citizens Hospital, Yokohama
- New Zealand (5):
  - North Shore Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
  - Tauranga Hospital, Tauranga
  - Wellington Regional Hospital (Ccdhb), Wellington
- Poland (5):
  - Pratia McM Krakow, Krakow
  - Wielospecjalistyczne Centrum Onkologii I Traumatologii Im M Kopernika W Lodzi, Lodz
  - Uniwersytecki Szpital Kliniczny Nr W Lublinie, Lublin
  - Aidport Sp Z O O, Skorzewo
  - Dolnoslaskie Centrum Onkologii, Pulmonologii I Hematologii, Wroclaw
- Auxilio Mutuo Cancer Center, San Juan, Puerto Rico
- South Korea (8):
  - Pusan National University Hospital, Seogu, Busan Gwang'yeogsi
  - Seoul National University Bundang Hospital, BundangGu SeongnamSi, Gyeonggi-do
  - Samsung Medical Center, GangnamGu, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St Marys Hospital, SeochoGu, Seoul Teugbyeolsi
  - Severance Hospital Yonsei University Health System, SeodaemunGu, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center, SongpaGu, Seoul Teugbyeolsi
  - The Catholic University of Korea, Yeouido St Marys Hospital, Yeongdeungpo-gu, Seoul Teugbyeolsi
- Spain (4):
  - Hospital Clinic de Barcelona, Barcelona
  - Ico H Duran I Reynals, Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - H Puerta de Hierro Majadahonda, Majadahonda
- Turkey (Türkiye) (3):
  - Etlik City Hospital, Ankara
  - Antalya Memorial Hospital, Dokuma
  - Kocaeli Universitesi Tip Fakultesi, Kocaeli
- United Kingdom (6):
  - The Royal Bournemouth and Christchurch Hospitals Nhs Foundation, Bournemouth
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Churchill Hospital Oxford University Hospital Nhs Trust, Headington
  - University College Hospital, London
  - Clatterbridge Cancer Centre, Metropolitan Borough of Wirral
  - Derriford Hospital, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
BeOne shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeOne shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeOne review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beonemedicines.com/science/clinical-trials/